CLINICAL TRIAL: NCT00241358
Title: A Phase I/II Study Evaluating the Safety and Efficacy of AMD3100 for the Mobilization and Transplantation of HLA-Matched Sibling Donor Hematopoietic Stem Cells in Patients With Advanced Hematological Malignancies
Brief Title: Study Evaluating AMD3100 for Transplantation of Sibling Donor Stem Cells in Patients With Hematological Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-0349
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic; Leukemia, Lymphoblastic, Acute; Lymphocytic Leukemia, Chronic; Myelodysplastic Syndromes; Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease
Keywords: Plerixafor; Stem cell transplantation; Stem cells; Mobilization
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Myelodysplastic Syndromes; Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — plerixafor; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Subcutaneous (SC) Treatment Plan - Donor (Active Comparator): * Day 1: Mobilization with 240 mcg/kg SC AMD3100 and leukopheresis
  * If PBSC collected are not adequate, then donor will again be mobilized with AMD3100 and have leukopheresis collection on day 3.
  Interventions: Drug: AMD3100
- Intravenous (IV) Treatment Plan - Donor (Experimental): * Day -3: Mobilization with 80-480 mcg/kg/day IV AMD3100 and PK analysis
  * Day 1: Mobilization with 240 mcg/kg/day SC AMD3100 and leukopheresis
  * If PBSC collected are not adequate, then donor will again be mobilized with AMD3100 and have leukopheresis collection on day 3.
  Interventions: Drug: AMD3100
- Recipients (Other): * Conditioning Regimen
    * Cyclophosphamide 60mg/kg/day on Days -3 and -2
    * TBI 550cGy on Day -1
  * GVHD prophylaxis
    *Cyclosporin 3.0mg/kg/day beginning on Day -1 then tapered through Day +100
  * PBSC transplant on Day 0
  Interventions: Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: AMD3100
  Other Names: Plerixafor
  Arms: Intravenous (IV) Treatment Plan - Donor; Subcutaneous (SC) Treatment Plan - Donor
Procedure: Stem Cell Transplant
  Arms: Recipients

SUMMARY:
The purpose of this study is to determine if peripheral blood cells collected following AMD3100 mobilization can be used safely for hematopoietic cell transplantation into HLA-matched recipients.

DETAILED DESCRIPTION:
This study will determine if peripheral blood cells collected following AMD3100 mobilization can be used safely for hematopoietic cell transplantation into HLA-matched recipients.

ELIGIBILITY:
Inclusion Criteria:

Donor criteria:

* Donor is 18 to 70 years of age inclusive
* If female and of child-bearing age, must be:

  * non-pregnant,
  * not breast feeding and
  * using adequate contraception
* Donor is a 6/6 HLA-matched sibling willing to donate peripheral blood stem cell for transplant
* Donor must be willing to provide written informed consent.
* Adequate cardiac function with no history of congestive heart failure and no history of atrial fibrillation or ventricular tachyarrhythmia.
* Adequate renal function as defined by a serum creatinine clearance of ≥75% of normal (Cockcroft-Gault equation)
* Adequate hepatic function as defined by a total bilirubin <2x normal or absence of hepatic fibrosis/cirrhosis
* Adequate neurologic function as defined by:

  * No evidence of a severe central or peripheral neurologic abnormality.
  * No history of cerebrovascular accident or seizure disorder requiring anticonvulsant medication
* Must be HIV-1 & 2 antibody, HIV-1 antigen, and HTLV-I & II antibody sero-negative, by FDA licensed test.
* Must have an ECOG performance status of 0 or 1
* Must demonstrate ability to be compliant with study regimen.
* Must not have an active infection at the time of study entry
* Not have active alcohol or substance abuse within 6 months of study entry
* Not currently enrolled in another investigational agent study
* Not have any medical condition, which, in the opinion of the clinical investigator, would interfere with his/her evaluation

Recipient criteria:

* 18 to 65 years of age inclusive
* Willing and has a 6/6 HLA-matched sibling willing to donate PBSC for transplant
* Provide signed informed consent
* If female and of child-bearing age, must be:

  * non-pregnant,
  * not breast feeding, and
  * using adequate contraception

Patient must have one of the following diagnoses:

* AML in 1st or subsequent remission or in relapse
* ALL in 1st or subsequent remission or in relapse
* MDS and intermediate 1 or 2, or high risk by the International Prognostic Scoring System
* CML in accelerated or second chronic phase
* NHL or HD in 2nd or greater complete remission, partial remission,or refractory relapse
* CLL Rai Stage 2-4, failing at least 2 prior regimens
* MM Stage 2-3
* Adequate cardiac function with a left ventricular ejection fraction ≥ 40%
* Adequate pulmonary function defined as:

  * No severe or symptomatic restrictive or obstructive lung disease, and
  * formal pulmonary function testing showing an forced expiratory volume at 1 second (FEV1) ≥50% of predicted and a diffusion capacity of the lung for carbon monoxide (DLCO) ≥40% of predicted, corrected for hemoglobin
* Adequate renal function as defined by a serum creatinine clearance of ≥75% of normal (Cockcroft-Gault equation)
* Adequate hepatic function as defined by a total bilirubin <2x normal or absence of hepatic fibrosis/cirrhosis
* Adequate neurologic function as defined by no evidence of a severe central or peripheral neurologic abnormality. Patients with a history of previous central nervous system tumor involvement are eligible provided they are without symptoms or signs and the CNS is now free of disease on lumbar puncture and CT scan of the brain
* No evidence of active infection at the time of the transplant preparative regimen or at the time of transplantation
* Patient must be HIV-1 & 2 antibody, HIV-1 antigen, and HTLV-I & II antibody sero-negative, by FDA licensed test
* ECOG performance status of 0 or 1
* Must demonstrate ability to be compliant with medical regimen
* Not have active alcohol or substance abuse within 6 months of study entry
* Not be concurrently enrolled on another study involving an investigational agent
* Not have any medical condition, which, in the opinion of the clinical investigator, would interfere with the evaluation of the patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2004-05; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F. DiPersio, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devine SM, Vij R, Rettig M, Todt L, McGlauchlen K, Fisher N, Devine H, Link DC, Calandra G, Bridger G, Westervelt P, Dipersio JF. Rapid mobilization of functional donor hematopoietic cells without G-CSF using AMD3100, an antagonist of the CXCR4/SDF-1 interaction. Blood. 2008 Aug 15;112(4):990-8. doi: 10.1182/blood-2007-12-130179. Epub 2008 Apr 21. PMID 18426988
- [Background] Devine SM, Flomenberg N, Vesole DH, Liesveld J, Weisdorf D, Badel K, Calandra G, DiPersio JF. Rapid mobilization of CD34+ cells following administration of the CXCR4 antagonist AMD3100 to patients with multiple myeloma and non-Hodgkin's lymphoma. J Clin Oncol. 2004 Mar 15;22(6):1095-102. doi: 10.1200/JCO.2004.07.131. PMID 15020611
- [Background] Flomenberg N, Devine SM, Dipersio JF, Liesveld JL, McCarty JM, Rowley SD, Vesole DH, Badel K, Calandra G. The use of AMD3100 plus G-CSF for autologous hematopoietic progenitor cell mobilization is superior to G-CSF alone. Blood. 2005 Sep 1;106(5):1867-74. doi: 10.1182/blood-2005-02-0468. Epub 2005 May 12. PMID 15890685
- [Derived] Schroeder MA, Rettig MP, Lopez S, Christ S, Fiala M, Eades W, Mir FA, Shao J, McFarland K, Trinkaus K, Shannon W, Deych E, Yu J, Vij R, Stockerl-Goldstein K, Cashen AF, Uy GL, Abboud CN, Westervelt P, DiPersio JF. Mobilization of allogeneic peripheral blood stem cell donors with intravenous plerixafor mobilizes a unique graft. Blood. 2017 May 11;129(19):2680-2692. doi: 10.1182/blood-2016-09-739722. Epub 2017 Mar 14. PMID 28292947
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was opened to participant enrollment on 05/14/2004 and closed to participant enrollment on 01/26/2009.
Period: Overall Study
Arm/Group | Subcutaneous (SC) Treatment Plan - Donor | Recipients | Intravenous (IV) Treatment Plan - Donor
Started | 25 | 46 | 21
Completed | 25 | 45 | 20
Not Completed | 0 | 1 | 1
Not completed — Determined to be not ineligible | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subcutaneous (SC) Treatment Plan - Donor | Recipients | Intravenous (IV) Treatment Plan - Donor | Total
Number analyzed (Participants) | 25 | 46 | 21 | 92
Age, Continuous [Median (Full Range); unit: years] | 54 [24 to 66] | 53 [23 to 66] | 51 [21 to 67] | 52 [21 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 26 | 8 | 39
  Male | 20 | 20 | 13 | 53
Region of Enrollment [Number; unit: participants]
  United States | 25 | 46 | 21 | 92

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Donors From Whom a Sufficient Number of Cells for Transplantation Are Collected in no More Than 2 LP Procedures Following Mobilization With AMD3100 (Donor Only)
Description: -Defined as the proportion of donors collecting >2.0x106 CD34+ cells/kg [recipient weight]
Time Frame: Day 1-3
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous (SC) Treatment Plan - Donor | Recipients | Intravenous (IV) Treatment Plan - Donor
Number analyzed (Participants) | 25 | 0 | 20
Participants | 22 |  | 19

2. Primary Outcome: Proportion of Recipients Who Experience Grade 2-4 Acute GVHD (Recipient Only)
Description: -Incidence and severity of acute GVHD (aGVHD) will be assessed based on the Seattle criteria
Time Frame: By Day 100 after transplant
Population: Only 38 recipients received stem cell products on study. The others were not eligible due to relapse/progression, poor donor collection, or receiving non-AMD3100 mobilized cells.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous (SC) Treatment Plan - Donor | Recipients | Intravenous (IV) Treatment Plan - Donor
Number analyzed (Participants) | 0 | 38 | 0
Participants |  | 15 |

3. Primary Outcome: Proportion of Recipients Who Successfully Engraft by Day +21 After Transplant (Recipient Only)
Description: -Defined as neutrophil count ≥ 500/ul following conditioning regimen induced nadir
Time Frame: Day +21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous (SC) Treatment Plan - Donor | Recipients | Intravenous (IV) Treatment Plan - Donor
Number analyzed (Participants) | 0 | 38 | 0
Participants |  | 37 |

4. Secondary Outcome: Proportion of Recipients Who Experience Chronic GVHD (Recipient Only)
Description: -Incidence and severity of chronic GVHD will be assessed based on the Seattle criteria
Time Frame: Between Day +100 and +365 post-transplant
Population: Only 28 recipients received stem cell products on study. The others were not eligible due to relapse/progression, poor donor collection, receiving non-AMD3100 mobilized cells, or death before day +100.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous (SC) Treatment Plan - Donor | Recipients | Intravenous (IV) Treatment Plan - Donor
Number analyzed (Participants) | 0 | 28 | 0
Participants |  | 10 |

5. Secondary Outcome: Proportion of Recipients Who Experience Mortality Before Day 100 After Transplant (Recipient Only)
Description: -Death that results from a transplant procedure related complication (e.g. infection, organ failure, hemorrhage, GVHD) rather than from relapse of the underlying disease or an unrelated cause
Time Frame: 100 days after transplant
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous (SC) Treatment Plan - Donor | Recipients | Intravenous (IV) Treatment Plan - Donor
Number analyzed (Participants) | 0 | 38 | 0
Participants |  | 2 |

6. Secondary Outcome: Quality of Life During Stem Cell Mobilization (Recipients Only)
Time Frame: 48-72 hours after last dose of AMD3100
Population: -Quality of life questionnaires were not collected from the recipients.
Arm/Group | Subcutaneous (SC) Treatment Plan - Donor | Recipients | Intravenous (IV) Treatment Plan - Donor
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Proportion of Donors Who Experience Infusional Toxicity (Donor Only)
Description: -Defined as hypersensitivity reactions. Evaluated by physical exam, blood pressure, heart rate, respirations and temperature one hour prior to the infusion and then 15 minutes, 30 minutes, one hour, 2 hours, and 4 hours post-infusion
Time Frame: Day +1 to +3 (SC donor arm) and Day -3 to +3 (IV donor arm)
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous (SC) Treatment Plan - Donor | Recipients | Intravenous (IV) Treatment Plan - Donor
Number analyzed (Participants) | 25 | 0 | 20
Participants | 0 |  | 0

8. Secondary Outcome: To Determine the Pharmacokinetics of IV AMD3100 (IV Donor Arm Only) as Measured by Cmax
Description: -Blood for pharmacokinetics were drawn prior to infusion, 15 minutes after infusion, 30 minutes after infusion, 45 minutes after infusion, 1 hour after infusion, 2 hours after infusion, 4 hours after infusion, 6 hours after infusions, and 24 hours after infusion
Time Frame: 0 to 24 hours after dose of IV AMD3100
Population: Pharmacokinetics were not performed on 2 patients who were considered replacement patients.
Measure: Mean (Full Range); unit: ng/ml
Arm/Group | Subcutaneous (SC) Treatment Plan - Donor | Recipients | Intravenous (IV) Treatment Plan - Donor
Number analyzed (Participants) | 0 | 0 | 19
ng/ml |  |  | 1058 [214 to 2150]

9. Secondary Outcome: To Determine the Pharmacokinetics of IV AMD3100 (IV Donor Arm Only) as Measured by Mean AUC From Time 0 to Infinity
Description: as for outcome 8
Time Frame: 0 to 24 hours after dose of IV AMD3100
Population: Pharmacokinetics were not performed on 2 patients who were considered replacement patients.
Measure: Mean (Full Range); unit: ng*hr/mL
Arm/Group | Subcutaneous (SC) Treatment Plan - Donor | Recipients | Intravenous (IV) Treatment Plan - Donor
Number analyzed (Participants) | 0 | 0 | 19
ng*hr/mL |  |  | 5150 [1243 to 11019]

ADVERSE EVENTS:
Groups:
- Donors: AMD3100 SC 240 ug/kg/actual donor weight on Day 1 and possibly Day 3
- Recipients: Stem Cell Transplantation Day 0
Arm/Group | Donors | Recipients
Serious Adverse Events (participants affected / at risk) | 2/46 | 12/46
Other Adverse Events (participants affected / at risk) | 46/46 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donors (N=46) | Recipients (N=46)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Ankle pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
C. Difficile infection (Infections and infestations) | 0 | 1
Confusion (Nervous system disorders) | 0 | 2
Congestive heart failure (Cardiac disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death due to disease progression (General disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Edema - extremities (General disorders) | 0 | 1
Emesis (Gastrointestinal disorders) | 0 | 1
Erythemous rash (Skin and subcutaneous tissue disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Fever (General disorders) | 1 | 2
Generalized weakness (General disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased bilirubin (Investigations) | 0 | 1
Increased creatinine (Renal and urinary disorders) | 0 | 1
Iron deficiency (Blood and lymphatic system disorders) | 1 | 0
Mouth pain (Gastrointestinal disorders) | 0 | 1
Mucositis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pancytopenia (Investigations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 3
Sepsis (Infections and infestations) | 0 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 1
Vasovagal reaction (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Weight loss (Investigations) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donors (N=46) | Recipients (N=46)
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4
Anasarca (General disorders) | 0 | 3
Anemia (Blood and lymphatic system disorders) | 2 | 0
Ankle pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 7
Arm pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Bacteremia (Infections and infestations) | 0 | 3
Bladder spasm (Renal and urinary disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 3 | 4
Bronchospasm wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bruising (Skin and subcutaneous tissue disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Chills (General disorders) | 3 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Cold sensation (General disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 6
Confusion (Psychiatric disorders) | 0 | 2
Congestive heart failure (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Cramping (Gastrointestinal disorders) | 3 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 10 | 16
Distension/abdominal bloating (Gastrointestinal disorders) | 4 | 2
Dizziness (Nervous system disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 1
Edema/larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Extrapyramidal involuntary movement (Nervous system disorders) | 2 | 3
Extremity walking (gait/walking) (Musculoskeletal and connective tissue disorders) | 0 | 3
Facial edema (head and neck) (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 17
Febrile neutropenia (Infections and infestations) | 0 | 19
Feet tremor (Nervous system disorders) | 0 | 1
Fever (General disorders) | 0 | 6
Fistula, GI (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 8 | 0
Foliculitis (Infections and infestations) | 1 | 3
G-tube site infection (Infections and infestations) | 0 | 1
Generalized weakness (General disorders) | 0 | 4
Hand tremor (Nervous system disorders) | 0 | 6
Headache (Nervous system disorders) | 2 | 7
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 1
Hemoptisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Hyperbilirubinemia (Investigations) | 0 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Hypotension (Vascular disorders) | 3 | 0
Hypothermia (General disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 2
Injection site reaction (General disorders) | 9 | 0
Insomnia (Psychiatric disorders) | 1 | 2
Interstitial pneumonia (Infections and infestations) | 0 | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Knee pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Leg pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Lightheadedness (Nervous system disorders) | 13 | 0
Lower extremities edema (General disorders) | 0 | 4
Mental status change (Psychiatric disorders) | 0 | 2
Mood alteration (Psychiatric disorders) | 1 | 5
Mucositis (Gastrointestinal disorders) | 0 | 18
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 16
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-specific ST abnormality (Cardiac disorders) | 1 | 0
Otitis, middle ear (Ear and labyrinth disorders) | 0 | 1
Paranasal reactions (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Petequiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 14
Renal failure (Renal and urinary disorders) | 0 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Seizure (Nervous system disorders) | 0 | 3
Sensory neuropathy (Nervous system disorders) | 15 | 3
Shoulder blade pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Spine pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spine pain (Nervous system disorders) | 1 | 0
Sweating (diaphoresis) (General disorders) | 5 | 0
Tachycardia (Cardiac disorders) | 0 | 5
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Throat pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thrombosis/embolism (DVT) (Vascular disorders) | 2 | 3
U wave (Cardiac disorders) | 1 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 2
Urinary color change (Renal and urinary disorders) | 0 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 4
Vasovagal episode (Cardiac disorders) | 2 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Viremia (Infections and infestations) | 0 | 3
Vitreous hemorrhage (Eye disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 16
Warm sensation (General disorders) | 5 | 0
Watery eye (tearing) (Eye disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes